CLINICAL TRIAL: NCT06192927
Title: A Phase 2, Multi-Centre, Randomised, Double-Blind, Sham Controlled Proof of Concept Trial Evaluating the Efficacy and Safety of TenoMiR by Injection in Subjects With Lateral Epicondylitis
Brief Title: Efficacy and Safety of TenoMiR in Lateral Epicondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Causeway Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CWT-TE2
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TenoMiR intralesional injection (Experimental): Drug: TenoMiR (Low Dose), Single injection Mimic of miR29a
  Other Names:
  • CWT-001
  Drug: TenoMiR (High Dose), Single injection Mimic of miR29a
  Other Names:
  • CWT-001
  Interventions: Drug: TenoMiR
- 0.9% saline subcutaneous sham injection (Sham Comparator): Drug: 0.9% saline Subcutaneous single injection
  Interventions: Drug: 0.9% Sodium Chloride Injection

INTERVENTIONS:
Drug: TenoMiR — Single intralesional injection
  Other Names: CWT-001
  Arms: TenoMiR intralesional injection
Drug: 0.9% Sodium Chloride Injection — Single subcutaneous injection
  Arms: 0.9% saline subcutaneous sham injection

SUMMARY:
This study is testing a drug called TenoMiR that is being developed for the treatment of tennis elbow (lateral epicondylitis). The study drug is a new compound that works by improving the quality of the collagen which helps repair damage to the elbow. The study drug is being developed in the hope of providing a more reliable treatment than those currently available and can be given at the time of first diagnosis, so that recovery can begin as soon as possible. The study drug has been tested in humans in an earlier study, and appeared to be safe and well-tolerated. This study aims to test the study drug in a larger number of participants.

DETAILED DESCRIPTION:
TenoMiR a chemically synthesised mimic of microRNA-29a (miR29a) which has improved stability, activity and cellular uptake while being non-immunogenic, has been created to restore miR29a levels back to pre-injury levels. TenoMiR is unique in directly targeting the key changes in collagen production associated with tendinopathy. Unlike other therapies, TenoMiR has a well-defined mode-of-action that is supported by a wealth of scientific data.

Moreover, treatment with TenoMiR does not require invasive biopsies and can be delivered at the point of initial diagnosis initiating recovery at the very earliest time. This is a global multicentre study which will test TenoMiR in a larger population, to follow on from the previous Phase 1b study in which TenoMiR appeared to be both safe and well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria.

1. Subject has a clinical diagnosis of lateral epicondylitis.
2. Aside from lateral epicondylitis, the subject is otherwise healthy as determined by a responsible physician, based on medical history, physical examinations, concomitant medication, vital signs, 12-lead ECGs and clinical laboratory evaluations. Laboratory values may be retested once at the discretion of the Investigator.
3. Subject's symptoms can be reproduced with resisted supination or wrist dorsiflexion (as confirmed by tenderness at lateral epicondyle and positive pick up back of chair sign).
4. Subject's symptoms have persisted for at least 6 weeks to 9 months, despite conservative treatment that includes 1 or combinations of:

   1. Physical therapy
   2. Splinting
   3. NSAIDs

Exclusion Criteria:

Subjects with any of the following will be excluded from study participation:

1. Subject has undergone previous corticosteroid injection therapy to the affected elbow in less than 6 months prior to enrolment.
2. Subjects unwilling or unable to discontinue use of pain medication (opiate or NSAID) from at least 1 week prior to Investigational Medicinal Product (IMP) administration.
3. Subject has received previous Platelet-Rich Plasma (PRP) injection to the affected elbow.
4. Subject uses or has recent use of medications known to affect the skeleton (e.g., glucocorticoid usage >5 mg/day, fluoroquinolone antibiotics).
5. Subject has undergone surgical intervention to the affected elbow for the treatment of lateral epicondylitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) pain score. Minimum score 0 (no pain), Maximum score 10 (worst possible pain) | 90 days
  Changes in pain score per group

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder, and Hand (QuickDASH) score. Minimum score 0 (no disability), Maximum score 100 (most severe disability) | 90 days
  Changes in QuickDASH per group
Patient Rated Tennis Elbow Evaluation (PRTEE) score. Minimum Score 0 (no pain or disability) Maximum Score 100 (worst pain and disability) | 90 days
  Changes in PRTEE per group
American Shoulder and Elbow Surgeons Elbow (ASES-E) score. Minimum score 0 (no pain or disability), Maximum score 144 (worst pain or disability) | 90 days
  Changes in ASES-E per group
Ultrasound assessment | 90 days
  Change in analysis of focal hypoechoic areas within the tendon per group. Evaluation will performed using a standardized scoring form (0=normal tendon, 1= mild tendinopathy, 2=moderate tendinopathy and 3= severe tendinopathy). Echogenicity will be characterized as hypoechogenic, normal, or hyperechogenic. Swelling (present or not present) of the tendon itself will be evaluated. Tendon thickness in mm will be noted. Calcifications (present or not present) will be assessed.
Ultrasound Tissue Characterisation (UTC) | 90 days
  Change in analysis of collagen echotypes within the tendon per group. Evaluation will be performed using the UTC system to objectively quantify greyscale tendon matrix changes into 4 different echotypes related to tendon integrity. Types I and II represent an organised matrix; Types III and IV represent a disorganised matrix. The composition of the tendon between groups will be assessed using the 4 listed echotypes. In addition, change between groups will be assessed by 3-dimensional ultrasound image of the tendon using standardised parameters (transducer tilt angle, depth and gain settings).
Incidence of Treatment-Emergent Adverse Events (AEs) between TenoMiR and sham comparator | 90 days
  Comparison of safety data between groups
Single dose pharmacokinetics (PK) of TenoMiR administration in subjects with lateral epicondylitis (Cmax). | 90 days
  Plasma PK by maximum drug plasma concentration (Cmax).

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Stanford Medicine, Redwood City, California
  - Hospital for Special Surgery, New York, New York
  - NYU Langone Health, New York, New York
- United Kingdom (6):
  - Panthera Biopartners, Enfield
  - Panthera Biopartners, Glasgow
  - Glasgow Clinical Research Facility, Glasgow
  - Panthera Biopartners, Preston
  - Panthera Biopartners, Rochdale
  - Panthera Biopartners, Sheffield